CLINICAL TRIAL: NCT03846193
Title: FOCUS: An Open Label First in Human Phase I/II Multicentre Study to Evaluate the Safety, Dose Response and Efficacy of GT005 Administered as a Single Subretinal Injection in Subjects With Macular Atrophy Due to AMD
Brief Title: FOCUS: A Phase I/II First in Human Study to Evaluate the Safety and Efficacy of GT005 Administered in Subjects With Dry AMD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to the interim analysis demonstrating lack of treatment efficacy.
Sponsor: Gyroscope Therapeutics Limited (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GT005-01; CPPY988A12101 (Other: Novartis)
Record Dates: First submitted 2019-02-13; First posted 2019-02-19 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Dry Age-related Macular Degeneration; Macular Degeneration; Retinal Disease; Eye Diseases; Retinal Degeneration; Geographic Atrophy; Macular Atrophy
Keywords: Dry Age-related Macular Degeneration (Dry AMD); AMD; Atrophic AMD; Geographic Atrophy (GA); Dry-AMD; Dry AMD
MeSH Terms: conditions — Macular Degeneration; Retinal Diseases; Eye Diseases; Retinal Degeneration; Geographic Atrophy; Anetoderma

STUDY DESIGN:
Intervention Model Description: A dose escalation study of the safety and efficacy of a single subretinal injection of GT005 in subjects with Macular Atrophy due to AMD
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- GT005 2E10 vg via Transvitreal Procedure (Experimental): GT005 2E10 vg via Transvitreal Procedure
  Interventions: Biological: GT005
- GT005 5E10 vg via Transvitreal Procedure (Experimental): GT005 5E10 vg via Transvitreal Procedure
  Interventions: Biological: GT005
- GT005 2E11 vg via Transvitreal Procedure (Experimental): GT005 2E11 vg via Transvitreal Procedure
  Interventions: Biological: GT005
- GT005 5E10 vg with Orbit Subretinal Delivery System (Experimental): GT005 5E10 vg with Orbit Subretinal Delivery System
  Interventions: Device: GT005 / Device: Orbit™ Subretinal Delivery System
- GT005 2E11 vg with Orbit Subretinal Delivery System (Experimental): GT005 2E11 vg with Orbit Subretinal Delivery System
  Interventions: Device: GT005 / Device: Orbit™ Subretinal Delivery System

INTERVENTIONS:
Biological: GT005 — GT005 is a recombinant, non-replicating AAV2 expressing human complement factor I (CFI). GT005 was administered as a single time subretinal injection into the study eye of subjects allocated to one of the two GT005 doses.
  Arms: GT005 2E10 vg via Transvitreal Procedure; GT005 2E11 vg via Transvitreal Procedure; GT005 5E10 vg via Transvitreal Procedure
Device: GT005 / Device: Orbit™ Subretinal Delivery System — GT005 is a recombinant, non-replicating AAV2 expressing human complement factor I (CFI).
  A single dose of GT005 was administered with subretinal injection via suprachoroidal cannulation approach.
  Device: Orbit™ Subretinal Delivery System
  Arms: GT005 2E11 vg with Orbit Subretinal Delivery System; GT005 5E10 vg with Orbit Subretinal Delivery System

SUMMARY:
This was an open label first in human Phase I/II multicentre study of GT005 in subjects with Macular Atrophy due to Age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
This was an open label first-in-human Phase I/II multicenter study to evaluate the safety, dose response and efficacy of GT005 in participants with Geographic atrophy (GA) due to Age-related macular degeneration (AMD).

The study treatment GT005 consists of an Adeno-associated virus serotype 2 (AAV2) expressing human complement factor I (hCFI). The treatment was administered as a single subretinal administration in one eye - the "study eye". Both eyes were assessed at the screening visit. If both eyes meet the eligibility criteria, the study eye will be the worse seeing eye, or the eye with the largest geographic atrophy (GA) lesion area for eyes with equivalent visual acuity, unless the participant (in consultation with the surgeon) expresses an alternative preference.

The study was conducted in 4 parts: in Part 1 and Part 2 GT005 was administered subretinally via transvitreal procedure; in Part 3 and 4 GT005 was delivered subretinally via a suprachoroidal cannulation with the Orbit Subretinal delivery system (SDS). The Orbit SDS is a 510(k) cleared device in the US, whereby Parts 3 and 4 were only conducted at US sites. The treatment consisted in 3 dose levels: low dose, 2E10 vector genomes (vg); medium dose, 5E10 vg; and high dose, 2E11 vg.

The study consisted of up to 13 visits over a 5-year period. All participants were assessed for the occurrence of treatment emergent adverse events (AE)s at each visit and underwent visual function and retinal imaging assessments and biological sampling as per the schedule of assessments.

This study was conducted in compliance with Independent ethics committees (IECs) / Institutional review boards (IRBs), informed consent regulations, the Declaration of Helsinki, nternational Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) Good Clinical Practice (GCP) Guidelines, and the Food and Drug Administration (FDA) guidance.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give consent to study participation
2. Have a clinical diagnosis of GA secondary to AMD in the study eye, as determined by the Investigator, and a diagnosis of AMD in the contralateral eye (except if the subject is monocular)
3. Cohorts 1 to 6: GA lesion(s) total size in the study eye must be ≥1.25mm2 and ≤17.5mm2.

   Cohort 7: GA lesion(s) total size in the study eye must be ≥1.25mm2
4. GA lesion(s) in the study eye must reside completely within the FAF fundus image
5. Cohorts 1 to 3: BCVA of ≤50 letters (6/36 Snellen acuity equivalent or worse) using ETDRS charts in the study eye Cohorts 4 to 7: BCVA of ≥24 letters (6/95 and 20/320 Snellen acuity equivalent or better) using ETDRS charts in the study eye
6. Aged ≥55 years
7. Able to attend all study visits and complete the study procedures
8. Women of child-bearing potential need to have a negative urine pregnancy test within two weeks prior to receiving the drug. A pregnancy test is not required for postmenopausal women (defined as being at least 12 consecutive months without menses) or those surgically sterilised (those having a bilateral tubal ligation/bilateral salpingectomy, bilateral tubal occlusive procedure, hysterectomy, or bilateral oophorectomy)

Exclusion Criteria:

1. Have evidence or history of Choroidal Neovascularisation (CNV) in the study eye. Subjects are permitted to have CNV in the fellow eye defined as either:

   1. Non-exudative/sub-clinical fellow eye CNV identified at screening, or
   2. Known history of fellow eye CNV with either ≥2 years since diagnosis or with no active treatment required in 6 months prior to screening
2. Presence of moderate/severe non-proliferative diabetic retinopathy or worse in the study eye
3. Have history of vitrectomy, sub-macular surgery, or macular photocoagulation in the study eye
4. History of intraocular surgery in the study eye within 12 weeks prior to Screening (Visit 1). Yttrium aluminum garnet capsulotomy is permitted if performed >10 weeks prior to Visit 1
5. Have clinically significant cataract that may require surgery during the study period in the study eye
6. Presence of moderate to severe glaucomatous optic neuropathy in the study eye; uncontrolled IOP despite the use of more than two topical agents; a history of glaucoma-filtering or valve surgery is also excluded
7. Axial myopia of greater than -8 diopters in the study eye
8. Have received any investigational product for the treatment of GA within the past 6 months or 5 half-lives (whichever is longer), other than nutritional supplements such as the Age-Related Eye Disease Study (AREDS) formula
9. Have received a gene or cell therapy at any time
10. Have a contraindication to the specified protocol corticosteroid regimen
11. Are unwilling to use two forms of contraception (one of which being a barrier method) for 90 days post-dosing, if relevant
12. Active malignancy within the past 12 months, except for: Appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or prostate cancer with a stable prostate-specific antigen (PSA) ≥12 months
13. Have any other significant ocular or non-ocular medical or psychiatric condition which, in the opinion of the Investigator, may either put the subject at risk or may influence the results of the study
14. Cohorts 5 to 7 only: presence of metallic objects or implanted stimulator devices in or near the head, including cochlear implants, deep brain stimulators, vagus nerve stimulators, and other implanted electrodes or stimulators

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Novartis Pharmaceuticals
Locations (13):
- United States (7):
  - Midwest Eye Institute, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Ophthalamic Consultants of Boston (OCB), Boston, Massachusetts
  - Pepose Vision Institute, Chesterfield, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Mid-Atlantic Retina, Philadelphia, Pennsylvania
- United Kingdom (6):
  - Bristol Eye Hospital, Bristol
  - Retina Clinic London, London
  - Moorfields Eye Hospital, London
  - Manchester Eye Hospital, Manchester
  - Oxford University Hospital, Oxford
  - Sunderland Eye Infirmary, Sunderland

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Dreismann AK, McClements ME, Barnard AR, Orhan E, Hughes JP, Lachmann PJ, MacLaren RE. Functional expression of complement factor I following AAV-mediated gene delivery in the retina of mice and human cells. Gene Ther. 2021 May;28(5):265-276. doi: 10.1038/s41434-021-00239-9. Epub 2021 Mar 10. PMID 33750925
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2646
- See also: Novartis Clinical Trial Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18286

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The delivery was attempted in 28 pts but was only successful in 25 pts. Of 3 pts where the GT005 delivery via Orbit SDS arms was not successful, 2 were treated via the transvitreal procedure, and 1 was disc. from treatment. (For 1 of the 3 pts, BSS delivery was successful, but not GT005 delivery.)
Period: Overall Study
Arm/Group | GT005 2E10 vg Via Transvitreal Procedure | GT005 5E10 vg Via Transvitreal Procedure | GT005 2E11 vg Via Transvitreal Procedure | GT005 5E10 vg With Orbit Subretinal Delivery System | GT005 2E11 vg With Orbit Subretinal Delivery System
Started | 6 | 10 | 15 | 5 | 22
Initially Randomized to Receive PPY988 With the Transvitreal Procedure | 4 | 10 | 15 | 0 | 0
Received PPY988 With the Transvitreal Procedure, After the Orbit-SDS Was Attempted Unsuccessfully (Received PPY988 with the Transvitreal Procedure, after the Orbit Subretinal Delivery System was attempted unsuccessfully (regardless if completed or disc early)) | 2 | 0 | 0 | 0 | 0
Initially Randomized to Receive PPY988 With the Orbit Subretinal Delivery System (Initially randomized to receive PPY988 with the Orbit Subretinal Delivery System (regardless if successful or unsuccessful)) | 0 | 0 | 0 | 5 | 22
Initially Randomized to Receive PPY988 With the Orbit Subretinal Delivery System (Initially randomized to receive PPY988 with the Orbit Subretinal Delivery System but the delivery was unsuccessful) | 1 | 0 | 0 | 2 | 0
Received PPY988 With the Transvitreal Procedure | 6 | 10 | 15 | 0 | 0
Received PPY988 With the Orbit Subretinal Delivery System | 0 | 0 | 0 | 3 | 22
Completed | 6 | 10 | 14 | 3 | 21
Not Completed | 0 | 0 | 1 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — switched to the GT005 2E10 vg via Transvitreal Procedure | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GT005 2E10 vg Via Transvitreal Procedure | GT005 5E10 vg Via Transvitreal Procedure | GT005 2E11 vg Via Transvitreal Procedure | GT005 5E10 vg With Orbit Subretinal Delivery System | GT005 2E11 vg With Orbit Subretinal Delivery System | Total
Number analyzed (Participants) | 6 | 10 | 15 | 3 | 22 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 81.7 (8.21) | 79.0 (5.12) | 80.5 (4.02) | 75.7 (4.73) | 77.3 (6.60) | 78.9 (5.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11 | 3 | 14 | 39
  Male | 1 | 4 | 4 | 0 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 10 | 14 | 3 | 22 | 55
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Ocular Treatment Emergent Adverse Events by Primary System Organ Class and Preferred Term for the Study Eye
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject.
  A TEAE is defined as any AE that develops after randomization or any AE already present that worsens following randomization. The primary summaries of AEs are based on TEAEs.
  System organ classes are sorted alphabetically, and preferred terms are sorted by decreasing overall frequency within system organ class.
Time Frame: Adverse events are reported from the single dose of study medication administration until end of study treatment plus 240 weeks post treatment, up to a maximum timeframe of approximately 240 weeks.
Population: Safety Analysis Set - All treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | GT005 2E10 vg Via Transvitreal Procedure | GT005 5E10 vg Via Transvitreal Procedure | GT005 2E11 vg Via Transvitreal Procedure | GT005 5E10 vg With Orbit Subretinal Delivery System | GT005 2E11 vg With Orbit Subretinal Delivery System
Number analyzed (Participants) | 6 | 10 | 15 | 3 | 22
Participants
  Subjects with at least one TEAE | 3 | 7 | 14 | 3 | 21
  Congenital, familial and genetic disorders | 0 | 0 | 1 | 0 | 0
  -Corneal dystrophy | 0 | 0 | 1 | 0 | 0
  Eye disorders | 3 | 6 | 13 | 3 | 21
  -Retinal pigmentation | 0 | 4 | 10 | 0 | 8
  -Conjunctival haemorrhage | 0 | 0 | 0 | 3 | 15
  -Cataract | 1 | 3 | 7 | 0 | 2
  -Retinal haemorrhage | 0 | 2 | 1 | 3 | 5
  -Dry eye | 1 | 2 | 2 | 0 | 2
  -Anterior chamber cell | 0 | 0 | 1 | 1 | 3
  -Retinal tear | 0 | 0 | 0 | 0 | 4
  -Blepharitis | 0 | 3 | 0 | 0 | 0
  -Conjunctival hyperaemia | 0 | 0 | 1 | 0 | 2
  -Neovascular age-related macular degeneration | 0 | 0 | 0 | 1 | 2
  -Visual field defect | 0 | 0 | 3 | 0 | 0
  -Charles Bonnet syndrome | 1 | 0 | 1 | 0 | 0
  -Eye pain | 0 | 0 | 1 | 0 | 1
  -Eyelid ptosis | 0 | 0 | 1 | 0 | 1
  -Visual acuity reduced | 1 | 0 | 0 | 0 | 1
  -Vitreous floaters | 0 | 0 | 1 | 1 | 0
  -Central vision loss | 0 | 0 | 1 | 0 | 0
  -Chalazion | 0 | 0 | 0 | 1 | 0
  -Choroidal haemorrhage | 0 | 0 | 0 | 0 | 1
  -Choroidal neovascularisation | 0 | 0 | 1 | 0 | 0
  -Conjunctival deposit | 0 | 0 | 0 | 0 | 1
  -Corneal oedema | 0 | 0 | 0 | 0 | 1
  -Dacryostenosis acquired | 0 | 1 | 0 | 0 | 0
  -Diplopia | 0 | 0 | 0 | 0 | 1
  -Eye discharge | 0 | 0 | 0 | 1 | 0
  -Eye pruritus | 0 | 1 | 0 | 0 | 0
  -Eyelid irritation | 0 | 0 | 0 | 1 | 0
  -Foreign body sensation in eyes | 0 | 0 | 0 | 0 | 1
  -Glaucoma | 0 | 0 | 0 | 0 | 1
  -Iridocyclitis | 0 | 0 | 1 | 0 | 0
  -Keratitis | 0 | 0 | 0 | 1 | 0
  -Macular hole | 0 | 0 | 1 | 0 | 0
  -Ocular discomfort | 0 | 0 | 0 | 0 | 1
  -Ocular hypertension | 0 | 1 | 0 | 0 | 0
  -Optic disc haemorrhage | 0 | 0 | 1 | 0 | 0
  -Periorbital oedema | 1 | 0 | 0 | 0 | 0
  -Posterior capsule opacification | 0 | 0 | 0 | 0 | 1
  -Retinal depigmentation | 0 | 0 | 0 | 0 | 1
  -Vision blurred | 0 | 0 | 1 | 0 | 0
  -Visual impairment | 0 | 0 | 1 | 0 | 0
  Infections and infestations | 0 | 3 | 0 | 0 | 2
  -Conjunctivitis | 0 | 0 | 0 | 0 | 2
  -Conjunctivitis viral | 0 | 2 | 0 | 0 | 0
  -Conjunctivitis bacterial | 0 | 1 | 0 | 0 | 0
  Injury, poisoning and procedural complications | 0 | 0 | 4 | 0 | 3
  -Procedural pain | 0 | 0 | 3 | 0 | 1
  -Corneal abrasion | 0 | 0 | 1 | 0 | 1
  -Post procedural discomfort | 0 | 0 | 0 | 0 | 1
  -Suture related complication | 0 | 0 | 1 | 0 | 0
  Investigations | 0 | 0 | 1 | 1 | 1
  -Intraocular pressure increased | 0 | 0 | 1 | 1 | 1
  Nervous system disorders | 0 | 0 | 0 | 1 | 0
  -Ophthalmic migraine | 0 | 0 | 0 | 1 | 0

2. Primary Outcome: Summary of Non-Ocular Treatment Emergent Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject.
  A TEAE is defined as any AE that develops after randomization or any AE already present that worsens following randomization. The primary summaries of AEs are based on TEAEs.
Time Frame: as for outcome 1
Population: Safety Analysis Set - All treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | GT005 2E10 vg Via Transvitreal Procedure | GT005 5E10 vg Via Transvitreal Procedure | GT005 2E11 vg Via Transvitreal Procedure | GT005 5E10 vg With Orbit Subretinal Delivery System | GT005 2E11 vg With Orbit Subretinal Delivery System
Number analyzed (Participants) | 6 | 10 | 15 | 3 | 22
Participants | 4 | 10 | 14 | 3 | 16

3. Primary Outcome: Summary of Ocular Serious Treatment-Emergent Adverse Events in the Study Eye by System Organ Class and Preferred
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Safety Analysis Set - All treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | GT005 2E10 vg Via Transvitreal Procedure | GT005 5E10 vg Via Transvitreal Procedure | GT005 2E11 vg Via Transvitreal Procedure | GT005 5E10 vg With Orbit Subretinal Delivery System | GT005 2E11 vg With Orbit Subretinal Delivery System
Number analyzed (Participants) | 6 | 10 | 15 | 3 | 22
Participants | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Best Corrected Visual Acuity (BCVA) (in Early Treatment Diabetic Retinopathy Study (ETDRS) Letters) in the Study Eye
Description: Best corrected visual acuity (BCVA) was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Min and max possible scores are 0-100 respectively. A higher score represents better visual functioning.
Time Frame: Up to Week 240
Population: Full Analysis Set - All treated patients with a valid measurement without a protocol deviation with impact
Measure: Mean (Standard Deviation); unit: ETDRS letters read
Arm/Group | GT005 2E10 vg Via Transvitreal Procedure | GT005 5E10 vg Via Transvitreal Procedure | GT005 2E11 vg Via Transvitreal Procedure | GT005 5E10 vg With Orbit Subretinal Delivery System | GT005 2E11 vg With Orbit Subretinal Delivery System
Number analyzed (Participants) | 6 | 10 | 15 | 3 | 22
ETDRS letters read
  Week 1 | 39.33 (16.145) | 47.20 (16.151) | 47.20 (17.449) | 62.00 (17.436) | 52.59 (15.822)
  Week 5 (n=6,10,14,3,22): number analyzed (Participants) | 6 | 10 | 14 | 3 | 22
  Week 5 (n=6,10,14,3,22) | 42.00 (20.258) | 46.90 (13.916) | 45.57 (19.747) | 62.67 (19.425) | 52.14 (18.838)
  Week 8 (n=3,4,6,3,21): number analyzed (Participants) | 3 | 4 | 6 | 3 | 21
  Week 8 (n=3,4,6,3,21) | 60.33 (9.074) | 55.25 (9.674) | 55.67 (12.675) | 65.33 (16.442) | 52.52 (18.101)
  Week 12 (n=6,10,11,3,22): number analyzed (Participants) | 6 | 10 | 11 | 3 | 22
  Week 12 (n=6,10,11,3,22) | 44.33 (21.153) | 46.00 (15.563) | 54.73 (16.032) | 66.67 (16.166) | 54.68 (17.705)
  Week 24 (n=6,10,13,3,21): number analyzed (Participants) | 6 | 10 | 13 | 3 | 21
  Week 24 (n=6,10,13,3,21) | 42.67 (24.262) | 44.60 (13.810) | 48.92 (20.056) | 66.67 (19.218) | 52.76 (18.144)
  Week 36 (n=6,6,15,3,21): number analyzed (Participants) | 6 | 6 | 15 | 3 | 21
  Week 36 (n=6,6,15,3,21) | 39.00 (21.790) | 53.17 (12.983) | 43.80 (20.640) | 65.00 (21.932) | 52.29 (18.078)
  Week 48 (n=5,9,14,3,21): number analyzed (Participants) | 5 | 9 | 14 | 3 | 21
  Week 48 (n=5,9,14,3,21) | 40.60 (19.204) | 47.22 (13.953) | 47.86 (16.176) | 64.00 (20.518) | 51.19 (19.577)
  Week 72 (n=3,8,14,3,18): number analyzed (Participants) | 3 | 8 | 14 | 3 | 18
  Week 72 (n=3,8,14,3,18) | 32.67 (20.744) | 46.63 (15.408) | 46.93 (13.658) | 57.33 (16.258) | 51.72 (18.162)
  Week 96 (n=4,8,14,3,18): number analyzed (Participants) | 4 | 8 | 14 | 3 | 18
  Week 96 (n=4,8,14,3,18) | 31.00 (21.494) | 44.13 (12.484) | 43.57 (18.110) | 64.67 (24.583) | 51.72 (19.393)
  Week 144 (n=2,6,10,3,2): number analyzed (Participants) | 2 | 6 | 10 | 3 | 2
  Week 144 (n=2,6,10,3,2) | 26.50 (28.991) | 42.50 (9.628) | 43.90 (17.515) | 64.00 (18.520) | 56.00 (2.828)
  Week 192 (n=2,3,7,0,0): number analyzed (Participants) | 2 | 3 | 7 | 0 | 0
  Week 192 (n=2,3,7,0,0) | 26.50 (19.092) | 35.33 (8.505) | 36.43 (15.404) |  |
  Week 240 (n=2,1,2,0,0): number analyzed (Participants) | 2 | 1 | 2 | 0 | 0
  Week 240 (n=2,1,2,0,0) | 25.50 (16.263) | 28.00 | 25.50 (7.778) |  |

5. Secondary Outcome: Low-Luminance Deficit Best Corrected Visual Acuity (BCVA-LLVA) (in Early Treatment Diabetic Retinopathy Study (ETDRS) Letters) in the Study Eye
Description: Low-Luminance Deficit best corrected visual acuity (BCVA-LLVA) was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Min and max possible scores are 0-100 respectively. A higher score represents better visual functioning.
Time Frame: Up to Week 240
Population: Full Analysis Set - All treated patients with a valid measurement without a protocol deviation with impact
Measure: Mean (Standard Deviation); unit: ETDRS letters read
Arm/Group | GT005 2E10 vg Via Transvitreal Procedure | GT005 5E10 vg Via Transvitreal Procedure | GT005 2E11 vg Via Transvitreal Procedure | GT005 5E10 vg With Orbit Subretinal Delivery System | GT005 2E11 vg With Orbit Subretinal Delivery System
Number analyzed (Participants) | 6 | 10 | 15 | 3 | 22
ETDRS letters read
  Week 12 (n=3,9,11,3,22): number analyzed (Participants) | 3 | 9 | 11 | 3 | 22
  Week 12 (n=3,9,11,3,22) | 40.00 (21.517) | 14.67 (17.951) | 18.91 (14.321) | 28.67 (17.214) | 24.82 (16.229)
  Week 24 (n=6,10,13,3,21): number analyzed (Participants) | 6 | 10 | 13 | 3 | 21
  Week 24 (n=6,10,13,3,21) | 32.25 (29.205) | 15.80 (15.061) | 17.23 (13.893) | 27.00 (20.952) | 22.52 (14.473)
  Week 36 (n=4,6,15,3,20): number analyzed (Participants) | 4 | 6 | 15 | 3 | 20
  Week 36 (n=4,6,15,3,20) | 26.75 (24.865) | 21.00 (14.656) | 15.07 (15.144) | 30.00 (30.806) | 20.10 (14.242)
  Week 48 (n=5,9,14,3,21): number analyzed (Participants) | 5 | 9 | 14 | 3 | 21
  Week 48 (n=5,9,14,3,21) | 19.60 (14.415) | 15.11 (13.968) | 17.36 (15.736) | 31.67 (24.194) | 18.48 (13.938)
  Week 72 (n=3,8,14,3,18): number analyzed (Participants) | 3 | 8 | 14 | 3 | 18
  Week 72 (n=3,8,14,3,18) | 20.33 (14.154) | 13.13 (9.538) | 15.36 (17.095) | 33.67 (25.007) | 21.22 (12.735)
  Week 96 (n=4,8,14,3,18): number analyzed (Participants) | 4 | 8 | 14 | 3 | 18
  Week 96 (n=4,8,14,3,18) | 16.25 (9.215) | 8.88 (4.643) | 13.07 (15.711) | 36.00 (23.065) | 21.56 (13.984)
  Week 144 (n=2,6,10,3,2): number analyzed (Participants) | 2 | 6 | 10 | 3 | 2
  Week 144 (n=2,6,10,3,2) | 5.50 (6.364) | 6.50 (4.550) | 18.80 (18.760) | 39.67 (22.679) | 26.00 (26.870)
  Week 192 (n=2,3,7,0,0): number analyzed (Participants) | 2 | 3 | 7 | 0 | 0
  Week 192 (n=2,3,7,0,0) | 2.00 (1.414) | 5.00 (1.414) | 13.00 (9.220) |  |
  Week 240 (n=2,1,2,0,0): number analyzed (Participants) | 2 | 1 | 2 | 0 | 0
  Week 240 (n=2,1,2,0,0) | 7.50 (2.121) | 9.00 | 5.50 (3.536) |  |

6. Secondary Outcome: Macular Sensitivity Parameters by Mesopic Microperimetry (MP) Over Time in the Study Eye - MP Bivariate Contour Ellipse Area (BCEA) 63 Area (deg2)
Description: Macular sensitivity as assessed by mesopic Microperimetry.
  Mesopic Microperimetry (MP) Bivariate contour ellipse area (BCEA) 63 Area.
Time Frame: Up to Week 240
Population: Full Analysis Set - All treated patients with a valid measurement without a protocol deviation with impact
Measure: Mean (Standard Deviation); unit: degrees squared (deg2)
Arm/Group | GT005 2E10 vg Via Transvitreal Procedure | GT005 5E10 vg Via Transvitreal Procedure | GT005 2E11 vg Via Transvitreal Procedure | GT005 5E10 vg With Orbit Subretinal Delivery System | GT005 2E11 vg With Orbit Subretinal Delivery System
Number analyzed (Participants) | 3 | 9 | 14 | 3 | 11
degrees squared (deg2)
  Week 12 (n=2,9,11,1,10): number analyzed (Participants) | 2 | 9 | 11 | 1 | 10
  Week 12 (n=2,9,11,1,10) | 16.80 (5.940) | 15.64 (13.013) | 7.82 (8.232) | 36.90 | 5.97 (3.726)
  Week 24 (n=3,9,10,3,11): number analyzed (Participants) | 3 | 9 | 10 | 3 | 11
  Week 24 (n=3,9,10,3,11) | 16.17 (15.970) | 17.10 (17.891) | 12.13 (11.483) | 14.40 (20.809) | 10.38 (11.050)
  Week 48 (n=2,9,14,2,10): number analyzed (Participants) | 2 | 9 | 14 | 2 | 10
  Week 48 (n=2,9,14,2,10) | 8.50 (3.677) | 19.41 (19.557) | 11.96 (7.939) | 48.55 (50.134) | 11.34 (7.527)
  Week 72 (n=1,8,13,2,10): number analyzed (Participants) | 1 | 8 | 13 | 2 | 10
  Week 72 (n=1,8,13,2,10) | 17.80 | 13.33 (6.887) | 12.10 (7.970) | 27.65 (38.254) | 9.66 (6.935)
  Week 96 (n=2,8,13,1,7): number analyzed (Participants) | 2 | 8 | 13 | 1 | 7
  Week 96 (n=2,8,13,1,7) | 10.90 (2.546) | 14.65 (10.059) | 10.40 (6.389) | 0.30 | 6.11 (4.171)
  Week 144 (n=1,5,8,2,0): number analyzed (Participants) | 1 | 5 | 8 | 2 | 0
  Week 144 (n=1,5,8,2,0) | 12.20 | 18.80 (18.404) | 13.05 (7.505) | 4.30 (5.233) |
  Week 192 (1,2,7,0,0): number analyzed (Participants) | 1 | 2 | 7 | 0 | 0
  Week 192 (1,2,7,0,0) | 38.90 | 7.70 (0.283) | 13.80 (8.565) |  |
  Week 240 (1,1,2,0,0): number analyzed (Participants) | 1 | 1 | 2 | 0 | 0
  Week 240 (1,1,2,0,0) | 40.20 | 11.10 | 18.85 (24.395) |  |

7. Secondary Outcome: Macular Sensitivity Parameters by Mesopic Microperimetry (MP) Over Time in the Study Eye - MP Bivariate Contour Ellipse Area (BCEA) 95 Area (deg2)
Description: Macular sensitivity as assessed by mesopic Microperimetry.
  Mesopic Microperimetry (MP) Bivariate contour ellipse area (BCEA) 95 Area.
Time Frame: Up to Week 240
Population: Full Analysis Set - All treated patients with a valid measurement without a protocol deviation with impact
Measure: Mean (Standard Deviation); unit: degrees squared (deg2)
Arm/Group | GT005 2E10 vg Via Transvitreal Procedure | GT005 5E10 vg Via Transvitreal Procedure | GT005 2E11 vg Via Transvitreal Procedure | GT005 5E10 vg With Orbit Subretinal Delivery System | GT005 2E11 vg With Orbit Subretinal Delivery System
Number analyzed (Participants) | 3 | 9 | 14 | 3 | 11
degrees squared (deg2)
  Week 12 (n=2,9,11,1,10): number analyzed (Participants) | 2 | 9 | 11 | 1 | 10
  Week 12 (n=2,9,11,1,10) | 50.40 (17.819) | 46.86 (39.037) | 23.43 (24.638) | 110.70 | 17.81 (11.120)
  Week 24 (n=3,9,10,3,11): number analyzed (Participants) | 3 | 9 | 10 | 3 | 11
  Week 24 (n=3,9,10,3,11) | 48.37 (47.853) | 51.20 (53.652) | 36.28 (34.454) | 43.23 (62.405) | 31.09 (33.157)
  Week 48 (n=2,9,14,2,10): number analyzed (Participants) | 2 | 9 | 14 | 2 | 10
  Week 48 (n=2,9,14,2,10) | 25.45 (10.960) | 58.17 (58.589) | 35.79 (23.804) | 145.40 (150.331) | 33.96 (22.632)
  Week 72 (n=1,8,13,2,10): number analyzed (Participants) | 1 | 8 | 13 | 2 | 10
  Week 72 (n=1,8,13,2,10) | 53.40 | 39.94 (20.603) | 36.28 (23.848) | 82.90 (114.693) | 28.90 (20.743)
  Week 96 (n=2,8,13,1,7): number analyzed (Participants) | 2 | 8 | 13 | 1 | 7
  Week 96 (n=2,8,13,1,7) | 32.70 (7.495) | 43.90 (30.123) | 31.15 (19.152) | 0.80 | 18.30 (12.563)
  Week 144 (n=1,5,8,2,0): number analyzed (Participants) | 1 | 5 | 8 | 2 | 0
  Week 144 (n=1,5,8,2,0) | 36.60 | 56.32 (55.119) | 39.13 (22.511) | 12.85 (15.768) |
  Week 192 (1,2,7,0,0): number analyzed (Participants) | 1 | 2 | 7 | 0 | 0
  Week 192 (1,2,7,0,0) | 116.40 | 23.15 (0.778) | 41.33 (25.644) |  |
  Week 240 (1,1,2,0,0): number analyzed (Participants) | 1 | 1 | 2 | 0 | 0
  Week 240 (1,1,2,0,0) | 120.40 | 33.40 | 56.60 (73.115) |  |

8. Secondary Outcome: Macular Sensitivity Parameters by Mesopic Microperimetry (MP) Over Time in the Study Eye - MP Mean Sensitivity Decibel (dB)
Description: Macular sensitivity as assessed by mesopic Microperimetry
Time Frame: Up to Week 240
Population: Full Analysis Set - All treated patients with a valid measurement without a protocol deviation with impact
Measure: Mean (Standard Deviation); unit: Decibel (dB)
Arm/Group | GT005 2E10 vg Via Transvitreal Procedure | GT005 5E10 vg Via Transvitreal Procedure | GT005 2E11 vg Via Transvitreal Procedure | GT005 5E10 vg With Orbit Subretinal Delivery System | GT005 2E11 vg With Orbit Subretinal Delivery System
Number analyzed (Participants) | 3 | 9 | 14 | 3 | 11
Decibel (dB)
  Week 12 (n=2,9,11,1,10): number analyzed (Participants) | 2 | 9 | 11 | 1 | 10
  Week 12 (n=2,9,11,1,10) | 14.30 (2.121) | 7.76 (5.536) | 11.92 (5.165) | 0.90 | 13.51 (3.350)
  Week 24 (n=3,9,10,3,11): number analyzed (Participants) | 3 | 9 | 10 | 3 | 11
  Week 24 (n=3,9,10,3,11) | 4.20 (3.704) | 7.31 (5.736) | 10.63 (5.263) | 9.17 (8.259) | 13.02 (4.125)
  Week 48 (n=2,9,14,2,10): number analyzed (Participants) | 2 | 9 | 14 | 2 | 10
  Week 48 (n=2,9,14,2,10) | 5.75 (0.354) | 6.71 (6.065) | 9.96 (4.726) | 10.50 (4.525) | 12.19 (5.096)
  Week 72 (n=1,8,13,2,10): number analyzed (Participants) | 1 | 8 | 13 | 2 | 10
  Week 72 (n=1,8,13,2,10) | 13.00 | 6.89 (6.163) | 8.93 (5.416) | 8.55 (3.748) | 11.80 (3.435)
  Week 96 (n=2,8,13,1,7): number analyzed (Participants) | 2 | 8 | 13 | 1 | 7
  Week 96 (n=2,8,13,1,7) | 8.70 (2.687) | 6.06 (6.283) | 8.54 (4.859) | 10.20 | 11.19 (4.245)
  Week 144 (n=1,5,8,2,0): number analyzed (Participants) | 1 | 5 | 8 | 2 | 0
  Week 144 (n=1,5,8,2,0) | 4.00 | 7.52 (6.222) | 9.58 (6.123) | 12.45 (4.313) |
  Week 192 (1,2,7,0,0): number analyzed (Participants) | 1 | 2 | 7 | 0 | 0
  Week 192 (1,2,7,0,0) | 3.90 | 6.45 (5.728) | 6.87 (6.145) |  |
  Week 240 (1,1,2,0,0): number analyzed (Participants) | 1 | 1 | 2 | 0 | 0
  Week 240 (1,1,2,0,0) | 1.40 | 1.70 | 7.85 (6.435) |  |

9. Secondary Outcome: Macular Sensitivity Parameters by Mesopic Microperimetry (MP) Over Time in the Study Eye - MP Number of Scotomatous Points
Description: Macular sensitivity as assessed by mesopic Microperimetry
Time Frame: Up to Week 240
Population: Full Analysis Set - All treated patients with a valid measurement without a protocol deviation with impact
Measure: Mean (Standard Deviation); unit: MP Number of Scotomatous Points
Arm/Group | GT005 2E10 vg Via Transvitreal Procedure | GT005 5E10 vg Via Transvitreal Procedure | GT005 2E11 vg Via Transvitreal Procedure | GT005 5E10 vg With Orbit Subretinal Delivery System | GT005 2E11 vg With Orbit Subretinal Delivery System
Number analyzed (Participants) | 3 | 9 | 14 | 3 | 11
MP Number of Scotomatous Points
  Week 12 (n=2,9,11,1,10): number analyzed (Participants) | 2 | 9 | 11 | 1 | 10
  Week 12 (n=2,9,11,1,10) | 6.0 (0.00) | 29.3 (13.13) | 20.4 (12.78) | 44.0 | 11.9 (4.75)
  Week 24 (n=3,9,10,3,11): number analyzed (Participants) | 3 | 9 | 10 | 3 | 11
  Week 24 (n=3,9,10,3,11) | 44.3 (14.01) | 30.8 (13.15) | 23.6 (12.76) | 21.0 (22.52) | 12.5 (5.87)
  Week 48 (n=2,9,14,2,10): number analyzed (Participants) | 2 | 9 | 14 | 2 | 10
  Week 48 (n=2,9,14,2,10) | 40.0 (1.41) | 34.2 (15.08) | 22.0 (11.73) | 16.5 (7.78) | 15.0 (7.77)
  Week 72 (n=1,8,13,2,10): number analyzed (Participants) | 1 | 8 | 13 | 2 | 10
  Week 72 (n=1,8,13,2,10) | 9.0 | 35.0 (15.07) | 24.7 (12.30) | 19.5 (9.19) | 15.9 (7.37)
  Week 96 (n=2,8,13,1,7): number analyzed (Participants) | 2 | 8 | 13 | 1 | 7
  Week 96 (n=2,8,13,1,7) | 26.0 (18.38) | 36.4 (16.09) | 27.5 (13.33) | 17.0 | 17.0 (4.86)
  Week 144 (n=1,5,8,2,0): number analyzed (Participants) | 1 | 5 | 8 | 2 | 0
  Week 144 (n=1,5,8,2,0) | 44.0 | 32.2 (16.93) | 27.6 (15.82) | 17.0 (9.90) |
  Week 192 (1,2,7,0,0): number analyzed (Participants) | 1 | 2 | 7 | 0 | 0
  Week 192 (1,2,7,0,0) | 40.0 | 37.0 (22.63) | 32.4 (18.12) |  |
  Week 240 (1,1,2,0,0): number analyzed (Participants) | 1 | 1 | 2 | 0 | 0
  Week 240 (1,1,2,0,0) | 46.0 | 50.0 | 33.0 (16.97) |  |

10. Secondary Outcome: Macular Sensitivity Parameters by Mesopic Microperimetry (MP) Over Time in the Study Eye - MP Percent Fixation Loss (%)
Description: Macular sensitivity as assessed by mesopic Microperimetry
Time Frame: Up to Week 240
Population: Full Analysis Set - All treated patients with a valid measurement without a protocol deviation with impact
Measure: Mean (Standard Deviation); unit: MP Percent Fixation Loss (%)
Arm/Group | GT005 2E10 vg Via Transvitreal Procedure | GT005 5E10 vg Via Transvitreal Procedure | GT005 2E11 vg Via Transvitreal Procedure | GT005 5E10 vg With Orbit Subretinal Delivery System | GT005 2E11 vg With Orbit Subretinal Delivery System
Number analyzed (Participants) | 3 | 9 | 14 | 3 | 11
MP Percent Fixation Loss (%)
  Week 12 (n=2,9,11,1,10): number analyzed (Participants) | 2 | 9 | 11 | 1 | 10
  Week 12 (n=2,9,11,1,10) | 4.0 (5.66) | 9.8 (13.92) | 6.9 (8.69) | 0.0 | 5.5 (7.11)
  Week 24 (n=3,9,10,3,11): number analyzed (Participants) | 3 | 9 | 10 | 3 | 11
  Week 24 (n=3,9,10,3,11) | 0.0 (0.00) | 9.3 (17.00) | 6.4 (9.00) | 0.0 (0.00) | 11.3 (8.60)
  Week 48 (n=2,9,14,2,10): number analyzed (Participants) | 2 | 9 | 14 | 2 | 10
  Week 48 (n=2,9,14,2,10) | 0.0 (0.00) | 3.8 (7.64) | 10.5 (23.45) | 0.0 (0.00) | 4.6 (6.19)
  Week 72 (n=1,8,13,2,10): number analyzed (Participants) | 1 | 8 | 13 | 2 | 10
  Week 72 (n=1,8,13,2,10) | 13.0 | 1.8 (4.95) | 12.0 (25.31) | 4.0 (5.66) | 6.2 (8.52)
  Week 96 (n=2,8,13,1,7): number analyzed (Participants) | 2 | 8 | 13 | 1 | 7
  Week 96 (n=2,8,13,1,7) | 8.5 (12.02) | 6.5 (9.65) | 10.3 (9.06) | 0.0 | 7.6 (11.07)
  Week 144 (n=1,5,8,2,0): number analyzed (Participants) | 1 | 5 | 8 | 2 | 0
  Week 144 (n=1,5,8,2,0) | 0.0 | 0.0 (0.00) | 4.4 (8.11) | 6.5 (9.19) |
  Week 192 (1,2,7,0,0): number analyzed (Participants) | 1 | 2 | 7 | 0 | 0
  Week 192 (1,2,7,0,0) | 0.0 | 0.0 (0.00) | 1.7 (5.38) |  |
  Week 240 (1,1,2,0,0): number analyzed (Participants) | 1 | 1 | 2 | 0 | 0
  Week 240 (1,1,2,0,0) | 0.0 | 0.0 | 0.0 (0.00) |  |

11. Secondary Outcome: Change From Baseline Over Time in Square Root of Geographic Atrophy Area Size (mm) Via FAF in the Study Eye
Description: Change from baseline in GA size as assessed by fundus autofluorescence
Time Frame: Up to Week 240
Population: Full Analysis Set - for patients with a valid measurement without a protocol deviation with impact
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | GT005 2E10 vg Via Transvitreal Procedure | GT005 5E10 vg Via Transvitreal Procedure | GT005 2E11 vg Via Transvitreal Procedure | GT005 5E10 vg With Orbit Subretinal Delivery System | GT005 2E11 vg With Orbit Subretinal Delivery System
Number analyzed (Participants) | 6 | 10 | 15 | 3 | 21
mm
  Week 5 (n=6,10,13,3,20): number analyzed (Participants) | 6 | 10 | 13 | 3 | 20
  Week 5 (n=6,10,13,3,20) | 0.06 (0.081) | 0.06 (0.028) | 0.06 (0.045) | 0.17 (0.147) | 0.08 (0.064)
  Week 12 (n=6,10,10,3,21): number analyzed (Participants) | 6 | 10 | 10 | 3 | 21
  Week 12 (n=6,10,10,3,21) | 0.13 (0.105) | 0.09 (0.037) | 0.12 (0.061) | 0.26 (0.223) | 0.15 (0.096)
  Week 24 (n=6,10,13,3,19): number analyzed (Participants) | 6 | 10 | 13 | 3 | 19
  Week 24 (n=6,10,13,3,19) | 0.20 (0.161) | 0.13 (0.053) | 0.22 (0.109) | 0.37 (0.296) | 0.22 (0.111)
  Week 36 (n=5,5,15,3,19): number analyzed (Participants) | 5 | 5 | 15 | 3 | 19
  Week 36 (n=5,5,15,3,19) | 0.38 (0.232) | 0.18 (0.098) | 0.25 (0.101) | 0.40 (0.310) | 0.29 (0.130)
  Week 48 (n=5,9,13,3,21): number analyzed (Participants) | 5 | 9 | 13 | 3 | 21
  Week 48 (n=5,9,13,3,21) | 0.57 (0.259) | 0.23 (0.105) | 0.30 (0.118) | 0.48 (0.384) | 0.35 (0.155)
  Week 72 (n=3,8,14,3,17): number analyzed (Participants) | 3 | 8 | 14 | 3 | 17
  Week 72 (n=3,8,14,3,17) | 0.57 (0.374) | 0.27 (0.090) | 0.43 (0.214) | 0.57 (0.425) | 0.50 (0.247)
  Week 96 (n=4,8,13,2,18): number analyzed (Participants) | 4 | 8 | 13 | 2 | 18
  Week 96 (n=4,8,13,2,18) | 0.59 (0.424) | 0.33 (0.113) | 0.54 (0.246) | 0.70 (0.822) | 0.60 (0.282)
  Week 144 (n=2,6,8,3,2): number analyzed (Participants) | 2 | 6 | 8 | 3 | 2
  Week 144 (n=2,6,8,3,2) | 0.62 (0.137) | 0.42 (0.081) | 0.77 (0.329) | 0.99 (0.790) | 0.98 (0.144)
  Week 192 (n=2,2,5,0,0): number analyzed (Participants) | 2 | 2 | 5 | 0 | 0
  Week 192 (n=2,2,5,0,0) | 0.89 (0.112) | 0.46 (0.042) | 0.89 (0.346) |  |
  Week 240 (n=2,0,2,0,0): number analyzed (Participants) | 2 | 0 | 2 | 0 | 0
  Week 240 (n=2,0,2,0,0) | 1.07 (0.216) |  | 1.07 (0.007) |  |

12. Secondary Outcome: Delivery of GT005 to the Subretinal Space - Rate of Successful Delivery, % (US Only) Via the Orbit Subretinal Delivery System (SDS) Device
Description: The rate of successful delivery is an evaluation limited to the administration performed using the Orbit Subretinal Delivery System (SDS) device, which is a 510(k) cleared device in the US.
  The rate of successful delivery of GT005 is the number of full doses delivered divided by number of Orbit devices used.
  This endpoint evaluates the surgical procedure with the Orbit device, and it is independent of the dose administered, as the volume of GT005 administered was consistent across all arms and cohorts.
  The delivery was attempted in 28 pts but was only successful in 25 pts. Of 3 pts where the GT005 delivery via Orbit SDS arms was not successful, 2 were treated via the transvitreal procedure, and 1 was disc. from treatment. (For 1 of the 3 pts, BSS delivery was successful, but not GT005 delivery.) In all other efficacy tables, these 2 pts who were treated via the transvitreal procedure are included in the 1 of the 3 Transvitreal Procedure arms and not 1 of the 2 Orbit SDS arms.
Time Frame: Day 1
Population: All Enrolled Set - For the 28 participants in the US where the Orbit Subretinal Delivery System was attempted.
  34 devices were used for 28 total pts - some deliveries took more than 1 attempt before the delivery was successful. If a delivery failed, a new attempt with a new device was conducted.
  The arms for this endpoint are combined per the SAP, because the endpoint is independent of the dose; only the attempted and successful delivery via the Orbit SDS device is of relevance.
Measure: Number; unit: percent of devices
Units Other Than Participants: Orbit devices
Groups:
- Total US Patients: Total US Patients
Arm/Group | Total US Patients
Number analyzed (Participants) | 28
Number analyzed (Orbit devices) | 34
percent of devices | 70.6

13. Secondary Outcome: Delivery of Balanced Salt Solution (BSS) or BSS PLUS (BSS+) to the Subretinal Space - Rate of Successful Delivery, % (US Only) Via the Orbit Subretinal Delivery System (SDS) Device
Description: The rate of successful delivery is an evaluation limited to the administration performed using the Orbit Subretinal Delivery System (SDS) device, which is a 510(k) cleared device in the US.
  The rate of successful delivery of BSS was the number of full doses delivered divided by number of Orbit devices used.
  This endpoint evaluates the surgical procedure with the Orbit device, and it is independent of the dose administered, as the volume of BSS administered was consistent across all arms and cohorts.
  The delivery was attempted in 28 pts but was only successful in 25 pts. Of 3 pts where the GT005 delivery via Orbit SDS arms was not successful, 2 were treated via the transvitreal procedure, and 1 was disc. from treatment. (For 1 of the 3 pts, BSS delivery was successful, but not GT005 delivery.) In all other efficacy tables, these 2 pts who were treated via the transvitreal procedure are included in the 1 of the 3 Transvitreal Procedure arms and not 1 of the 2 Orbit SDS arms.
Time Frame: Day 1
Population: as for outcome 12
Measure: Number; unit: percent of devices
Units Other Than Participants: Orbit devices
Arm/Group | Total US Patients
Number analyzed (Participants) | 28
Number analyzed (Orbit devices) | 34
percent of devices | 76.5

14. Secondary Outcome: Summary of Ocular Treatment-Emergent Adverse Events Related to Surgical Procedure in the Study Eye
Description: Subjects with device related AEs and SAEs after subretinal delivery with Orbit SDS.
  An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject.
  A TEAE is defined as any AE that develops after randomization or any AE already present that worsens following randomization. The primary summaries of AEs are based on TEAEs.
  System organ classes are sorted alphabetically, and preferred terms are sorted by decreasing overall frequency within system organ class.
Time Frame: Day 1
Population: Safety Analysis Set - All treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | GT005 2E10 vg Via Transvitreal Procedure | GT005 5E10 vg Via Transvitreal Procedure | GT005 2E11 vg Via Transvitreal Procedure | GT005 5E10 vg With Orbit Subretinal Delivery System | GT005 2E11 vg With Orbit Subretinal Delivery System
Number analyzed (Participants) | 6 | 10 | 15 | 3 | 22
Participants
  Subjects with at least one TEAE Related to Surgical Procedure | 2 | 4 | 9 | 3 | 20
  Eye disorders | 2 | 4 | 8 | 3 | 20
  -Conjunctival haemorrhage | 0 | 0 | 0 | 3 | 14
  -Cataract | 1 | 3 | 7 | 0 | 0
  -Retinal pigmentation | 0 | 2 | 2 | 0 | 6
  -Retinal haemorrhage | 0 | 1 | 1 | 3 | 3
  -Anterior chamber cell | 0 | 0 | 1 | 1 | 3
  -Conjunctival hyperaemia | 0 | 0 | 1 | 0 | 2
  -Retinal tear | 0 | 0 | 0 | 0 | 3
  -Vitreous floaters | 0 | 0 | 1 | 1 | 0
  -Choroidal haemorrhage | 0 | 0 | 0 | 0 | 1
  -Choroidal neovascularisation | 0 | 0 | 1 | 0 | 0
  -Corneal oedema | 0 | 0 | 0 | 0 | 1
  -Dry eye | 1 | 0 | 0 | 0 | 0
  -Eye discharge | 0 | 0 | 0 | 1 | 0
  -Eye pain | 0 | 0 | 0 | 0 | 1
  -Eye pruritus | 0 | 1 | 0 | 0 | 0
  -Foreign body sensation in eyes | 0 | 0 | 0 | 0 | 1
  -Iridocyclitis | 0 | 0 | 1 | 0 | 0
  -Keratitis | 0 | 0 | 0 | 1 | 0
  -Ocular discomfort | 0 | 0 | 0 | 0 | 1
  -Periorbital oedema | 1 | 0 | 0 | 0 | 0
  Injury, poisoning and procedural complications | 0 | 0 | 2 | 0 | 3
  -Corneal abrasion | 0 | 0 | 1 | 0 | 1
  -Post procedural discomfort | 0 | 0 | 0 | 0 | 1
  -Procedural pain | 0 | 0 | 0 | 0 | 1
  -Suture related complication | 0 | 0 | 1 | 0 | 0
  Investigations | 0 | 0 | 1 | 0 | 0
  -Intraocular pressure increased | 0 | 0 | 1 | 0 | 0

15. Secondary Outcome: Summary of Non-Ocular Treatment-Emergent Adverse Events Related to Surgical Procedure
Description: as for outcome 14
Time Frame: Day 1
Population: Safety Analysis Set - All treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | GT005 2E10 vg Via Transvitreal Procedure | GT005 5E10 vg Via Transvitreal Procedure | GT005 2E11 vg Via Transvitreal Procedure | GT005 5E10 vg With Orbit Subretinal Delivery System | GT005 2E11 vg With Orbit Subretinal Delivery System
Number analyzed (Participants) | 6 | 10 | 15 | 3 | 22
Participants | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Summary of Ocular Serious Treatment-Emergent Adverse Events Related to Surgical Procedure in the Study Eye
Description: as for outcome 14
Time Frame: Day 1
Population: Safety Analysis Set - All treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | GT005 2E10 vg Via Transvitreal Procedure | GT005 5E10 vg Via Transvitreal Procedure | GT005 2E11 vg Via Transvitreal Procedure | GT005 5E10 vg With Orbit Subretinal Delivery System | GT005 2E11 vg With Orbit Subretinal Delivery System
Number analyzed (Participants) | 6 | 10 | 15 | 3 | 22
Participants | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Summary of Non-Ocular Serious Treatment-Emergent Adverse Events Related to Surgical Procedure
Description: as for outcome 14
Time Frame: Day 1
Population: Safety Analysis Set - All treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | GT005 2E10 vg Via Transvitreal Procedure | GT005 5E10 vg Via Transvitreal Procedure | GT005 2E11 vg Via Transvitreal Procedure | GT005 5E10 vg With Orbit Subretinal Delivery System | GT005 2E11 vg With Orbit Subretinal Delivery System
Number analyzed (Participants) | 6 | 10 | 15 | 3 | 22
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events are reported from the single dose of study medication administration until end of study treatment plus 240 weeks post treatment, up to a maximum timeframe of approximately 240 weeks.
Groups:
- Overall: Overall
Arm/Group | GT005 2E10 vg Via Transvitreal Procedure | GT005 5E10 vg Via Transvitreal Procedure | GT005 2E11 vg Via Transvitreal Procedure | GT005 5E10 vg With Orbit Subretinal Delivery System | GT005 2E11 vg With Orbit Subretinal Delivery System | Overall
All-Cause Mortality (participants affected / at risk) | 1/6 | 3/10 | 0/15 | 0/3 | 0/22 | 4/56
Serious Adverse Events (participants affected / at risk) | 2/6 | 6/10 | 4/15 | 0/3 | 5/22 | 17/56
Other Adverse Events (participants affected / at risk) | 4/6 | 10/10 | 15/15 | 3/3 | 22/22 | 54/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GT005 2E10 vg Via Transvitreal Procedure (N=6) | GT005 5E10 vg Via Transvitreal Procedure (N=10) | GT005 2E11 vg Via Transvitreal Procedure (N=15) | GT005 5E10 vg With Orbit Subretinal Delivery System (N=3) | GT005 2E11 vg With Orbit Subretinal Delivery System (N=22) | Overall (N=56)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Lymphatic system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 2
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GT005 2E10 vg Via Transvitreal Procedure (N=6) | GT005 5E10 vg Via Transvitreal Procedure (N=10) | GT005 2E11 vg Via Transvitreal Procedure (N=15) | GT005 5E10 vg With Orbit Subretinal Delivery System (N=3) | GT005 2E11 vg With Orbit Subretinal Delivery System (N=22) | Overall (N=56)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 2
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Corneal dystrophy - Fellow eye (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 1
Corneal dystrophy - Study eye (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 1
Ear pruritus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 1
Anterior chamber cell - Study eye (Eye disorders) | 0 | 0 | 1 | 1 | 3 | 5
Blepharitis - Fellow eye (Eye disorders) | 0 | 3 | 0 | 0 | 0 | 3
Blepharitis - Study eye (Eye disorders) | 0 | 3 | 0 | 0 | 0 | 3
Cataract - Fellow eye (Eye disorders) | 1 | 1 | 2 | 0 | 2 | 6
Cataract - Study eye (Eye disorders) | 1 | 3 | 7 | 0 | 2 | 13
Central vision loss - Study eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Chalazion - Study eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
Charles Bonnet syndrome - Fellow eye (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 2
Charles Bonnet syndrome - Study eye (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 2
Choroidal haemorrhage - Study eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Choroidal neovascularisation - Fellow eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Choroidal neovascularisation - Study eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Conjunctival deposit - Study eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Conjunctival haemorrhage - Study eye (Eye disorders) | 0 | 0 | 0 | 3 | 15 | 18
Conjunctival hyperaemia - Study eye (Eye disorders) | 0 | 0 | 1 | 0 | 2 | 3
Corneal oedema - Study eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dacryostenosis acquired - Study eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
Diplopia - Fellow eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Diplopia - Study eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dry eye - Fellow eye (Eye disorders) | 0 | 2 | 2 | 0 | 1 | 5
Dry eye - Study eye (Eye disorders) | 1 | 2 | 2 | 0 | 2 | 7
Eye discharge - Study eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
Eye pain - Fellow eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Eye pain - Study eye (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 2
Eye pruritus - Study eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
Eyelid irritation - Study eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
Eyelid ptosis - Fellow eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Eyelid ptosis - Study eye (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 2
Foreign body sensation in eyes - Study eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Glaucoma - Fellow eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Glaucoma - Study eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Iridocyclitis - Study eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Keratitis - Study eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
Macular hole - Study eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Neovascular age-related macular degeneration - Fellow eye (Eye disorders) | 0 | 0 | 2 | 1 | 0 | 3
Neovascular age-related macular degeneration - Study eye (Eye disorders) | 0 | 0 | 0 | 1 | 2 | 3
Ocular discomfort - Study eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Ocular hypertension - Fellow eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
Ocular hypertension - Study eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
Optic disc haemorrhage - Fellow eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Optic disc haemorrhage - Study eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Periorbital oedema - Study eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1
Posterior capsule opacification - Fellow eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Posterior capsule opacification - Study eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Retinal aneurysm rupture - Fellow eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Retinal depigmentation - Study eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Retinal haemorrhage - Fellow eye (Eye disorders) | 0 | 0 | 1 | 0 | 2 | 3
Retinal haemorrhage - Study eye (Eye disorders) | 0 | 2 | 1 | 3 | 5 | 11
Retinal pigmentation - Fellow eye (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 2
Retinal pigmentation - Study eye (Eye disorders) | 0 | 4 | 10 | 0 | 8 | 22
Retinal tear - Study eye (Eye disorders) | 0 | 0 | 0 | 0 | 4 | 4
Vision blurred - Fellow eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Vision blurred - Study eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Visual acuity reduced - Fellow eye (Eye disorders) | 0 | 3 | 0 | 1 | 0 | 4
Visual acuity reduced - Study eye (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 2
Visual field defect - Fellow eye (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 2
Visual field defect - Study eye (Eye disorders) | 0 | 0 | 3 | 0 | 0 | 3
Visual impairment - Fellow eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Visual impairment - Study eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Vitreous floaters - Study eye (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 3
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 3
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 2
Oesophageal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hernia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 0 | 0 | 1 | 3
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Polyp (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Vessel puncture site bruise (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 2 | 2 | 0 | 5 | 9
Cellulitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 3
Conjunctivitis - Fellow eye (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Conjunctivitis - Study eye (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2
Conjunctivitis bacterial - Fellow eye (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Conjunctivitis bacterial - Study eye (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Conjunctivitis viral - Fellow eye (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 2
Conjunctivitis viral - Study eye (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 2
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Hordeolum - Fellow eye (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 2
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 3 | 1 | 0 | 0 | 4
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 2
Staphylococcal skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 4
Viral sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 1 | 4
Corneal abrasion - Study eye (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 2
Eye contusion - Fellow eye (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 2 | 2 | 0 | 0 | 7
Foreign body in eye - Fellow eye (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Post procedural discomfort - Study eye (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Procedural pain - Study eye (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 1 | 4
Scrotal haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0 | 3
Skin wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Suture related complication - Study eye (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Blood albumin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Blood folate decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Blood potassium increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1 | 1 | 1 | 0 | 3
Coronavirus test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Heart rate irregular (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Intraocular pressure increased - Fellow eye (Investigations) | 0 | 0 | 1 | 1 | 0 | 2
Intraocular pressure increased - Study eye (Investigations) | 0 | 0 | 1 | 1 | 1 | 3
Lipids increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Protein C increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Protein total decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 2 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 2
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Sweat gland tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cerebral artery thrombosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cluster headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Dementia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 2
Meralgia paraesthetica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Ophthalmic migraine - Fellow eye (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Ophthalmic migraine - Study eye (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Vertebral artery occlusion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 2
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 0 | 3
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Haemosiderin stain (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 1 | 0 | 2 | 5
Hypertensive emergency (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 2
Poor peripheral circulation (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
Vein disorder (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1
Venous hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT03846193/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT03846193/SAP_001.pdf